CLINICAL TRIAL: NCT05962944
Title: Remote Rapid On-site Evaluation (ROSE) for Head and Neck Fine Needle Aspirations (FNA)
Brief Title: Remote Rapid Onsite Evaluation (ROSE) for Head and Neck Fine Needle Aspirations (FNA)
Acronym: Remote ROSE
Status: Completed | Type: Observational
Sponsor: Royal Cornwall Hospitals Trust (Other)
Responsible Party: Sponsor
Other Study IDs: RoyalCornwallHT
Record Dates: First submitted 2022-07-29; First posted 2023-07-27 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Head and Neck Neoplasms
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cytology fine needle aspiration samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Laboratory testing: Slides reviewed in the laboratory to test the platform for suitability prior to involving patients
  Interventions: Device: Olympus Cellsens software
- Remote ROSE on the same site as the laboratory: The next phase will involve remote ROSE being performed on the same site as the laboratory in an ultrasound room located on the Royal Cornwall Hospitals Truro site.
  Interventions: Device: Olympus Cellsens software
- Remote ROSE at a site external to the laboratory: Phase 3 will involved remote ROSE being performed on a different site to the laboratory. The ultrasound room at The Royal Cornwall Hospital's Camborne and Redruth site.
  Interventions: Device: Olympus Cellsens software

INTERVENTIONS:
Device: Olympus Cellsens software — Olympus cellsens software will be used to visualise the cells and MS teams screen share will be used to send the live images in real time.
  Other Names: Microsoft teams

SUMMARY:
Rapid On-Site Evaluation (ROSE) of cytology FNA samples performed by a Pathologist or Biomedical Scientist is a real time morphological assessment of the sample in the clinical setting with the aim of acquiring all the diagnostic material in one appointment resulting in reduction in costs, improved patient care and reduced referral to treatment time.

It is not practical or possible for the ROSE team to be present in every location where an FNA is performed. Telecytology (TC) or remote ROSE is a digital form of ROSE which allows a biomedical scientist or pathologist working in a remote laboratory to review the cytology slides in real time, using microscope images fed from the location where the FNA procedure is being performed.

DETAILED DESCRIPTION:
The new faster diagnostic standards (FDS) alongside NICE guidance and the British association of Head and Neck Oncologists (BAHNO) guidelines, state that ROSE should be provided for all FNA's. It is not practical or possible for the ROSE team to be present in every location where an FNA is performed. Telecytology (TC) or remote ROSE is a digital form of ROSE which allows a biomedical scientist or pathologist working in a remote laboratory to review the cytology slides in real time, using microscope images fed from the location where the FNA procedure is being performed.

A trained a clinical imaging assistant (CIA) will prepare the slides and drive the microscope in the ultrasound room. Using the Olympus software Cellsens and the screen share option in Microsoft teams, the remote biomedical scientist / pathologist will be able to assess the sample in real time and provide both verbal and written methods of communication (relevant clinical information and instructions). An additional camera will allow visualisation of the slide preparation and residual material in real time to the scientist / pathologist performing the assessment.

This study will investigate whether ROSE can be performed remotely. This study will be based in the cytology department at the Royal Cornwall Hospital as part of a service improvement. Phase 2 will involve the use of the Tower Block ultrasound room located on the Royal Cornwall Hospitals Truro site and in phase 3 the ultrasound room at The Royal Cornwall Hospital's Camborne and Redruth site.

Patients between the ages of 18 and 90 years attending for an ultrasound guided fine needle aspiration of lesions in the head and neck and supraclavicular fossa nodes will be consented for remote ROSE to be performed over a 12-month period.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants > 18-90 years of age
* Participants attending for an ultrasound guided fine needle aspiration of lesions in the head and neck and supraclavicular fossa nodes.
* All ethnicity or socioeconomic grouping that require an US FNA at RCHT over the 12-month study period.
* Able and willing to consent to the study

Exclusion Criteria:

* Anyone <18 years of age
* Patients that do not require an FNA after the initial ultrasound
* Any participants considered vulnerable will not be included in the study.
* This study involves testing the concept of remote ROSE rather than direct impact on patient care needs related to ethical of communication issues. For practical considerations and to prevent unnecessary anxiety for patients who are unable to read the information sheets and provide consent, these patients will not be included in the study.
* Unable or unwilling to consent to the study

Ages: 18 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Participants attending for an ultrasound guided fine needle aspiration of lesions in the head and neck and supraclavicular fossa nodes.
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2022-10-25 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-07-24 (Actual)

PRIMARY OUTCOMES:
Rapid on site evaluation can be provided using telecytology | 12 months
  To robustly test the concept of remote rapid on site evaluation for head and neck.
  The Scientist performing the remote ROSE will record the assessment findings:
  * Inadequate sampling - Advise repeat sampling
  * Adequate sampling - Stop procedure.
  * Diagnostic sampling but more material required. - Advise repeat sampling
  * Diagnostic sampling and sufficient cell yield - Stop procedure These findings will be compared with the final diagnostic outcomes (Final report) issued by the laboratory. The overall effectiveness of remote ROSE will be compared against current practice for head and neck FNA in terms of adequacy and diagnostic yield. If over 80% of samples obtained with remote ROSE are deemed adequate and sufficient then the trial will be regarded as successful. This prevents the majority of patients having to return for additional appointments and procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Leonie Wheeldon, Principal Investigator — Royal Cornwall Hospital
Locations (1):
- Royal Cornwall Hospital, Truro, Cornwall, United Kingdom